CLINICAL TRIAL: NCT00900185
Title: Retrospective Analysis of Endostatin Genotype in Prostate Cancer Patients to Assess the Association of a Single Nucleotide Polymorphism (D104N) in Endostatin and Prostate Cancer
Brief Title: Study of a Polymorphism in Patients With Prostate Cancer
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Other Study IDs: CDR0000304552; NCI-03-C-0153; NU-98U2
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2007-02

CONDITIONS: Prostate Cancer
Keywords: recurrent prostate cancer; stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Polymerase Chain Reaction; Amplified Fragment Length Polymorphism Analysis

INTERVENTIONS:
Genetic: mutation analysis
Genetic: polymerase chain reaction
Genetic: polymorphism analysis

SUMMARY:
RATIONALE: Studying samples of blood from patients with cancer and from healthy participants in the laboratory may help doctors learn more about changes that may occur in DNA.

PURPOSE: This laboratory study is looking at blood samples from patients with prostate cancer and from healthy participants to identify a polymorphism that may help in the study of prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the incidence of the D104N COL18A1 polymorphism in patients with prostate cancer.

Secondary

* Determine the incidence of this polymorphism in African-American patients with prostate cancer.

OUTLINE: This is a retrospective, multicenter study.

DNA is extracted from preexisting serum samples and polymerase chain reaction is performed to determine the genotype pattern.

PROJECTED ACCRUAL: A total of 500 patients and 250 healthy participants will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of prostate cancer OR healthy participant
* Patient enrolled on an IRB-approved clinical trial at the National Cancer Institute or Northwestern University, including, but not limited to, any of the following:

  * NCI-99-C-0052
  * NCI-95-C-0178
  * NCI-00-C-003
  * NCI-00-C-0080

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 750 (Estimated)

PRIMARY OUTCOMES:
Frequency of D104N COL18A1 polymorphism in patients with prostate cancer and in healthy participants

SECONDARY OUTCOMES:
Frequency of D104N COL18A1 polymorphism in African-American patients with prostate cancer and in healthy participants

CONTACTS AND LOCATIONS:
Overall Officials: William D. Figg, PharmD, Study Chair — National Cancer Institute (NCI)

REFERENCES:
- [Result] Macpherson GR, Singh AS, Bennett CL, Venzon DJ, Liewehr DJ, Franks ME, Dahut WL, Kantoff PW, Price DK, Figg WD. Genotyping and functional analysis of the D104N variant of human endostatin. Cancer Biol Ther. 2004 Dec;3(12):1298-303. doi: 10.4161/cbt.3.12.1453. Epub 2004 Dec 16. PMID 15662127
- [Result] Price DK, Macpherson GR, Dahut W, et al.: A mutation in COL18A1 and the association with prostate cancer. [Abstract] American Association for Cancer Research: 94th Annual Meeting, 11-14th July 2003, Washington, D.C. 44: A-4054, 810, 2003.